CLINICAL TRIAL: NCT06919159
Title: Intratumoral Heterogeneity on [18F]PSMA-1007 and [18F]FDG PET/CT in Predicting Invasion and Prognosis of Primary Prostate Cancer
Brief Title: Intratumoral Heterogeneity on [18F]PSMA and [18F]FDG PET/CT in Predicting Invasion and Prognosis of Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Jiequn Yu (Other)
Responsible Party: Sponsor-Investigator, Jiequn Yu, resident doctor, First Hospital of China Medical University
Organization: First Hospital of China Medical University (Other)
Other Study IDs: [2020]388
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer (Diagnosis); Prostate-specific Membrane Antigen; Positron Emission Tomography (PET)
Keywords: Fluorine-18-fluorodeoxyglucose; Heterogeneity
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- double positive group: patients with one type of PSMA+/FDG+ homogeneous segment
  Interventions: Diagnostic Test: PSMA PET/CT scan; Diagnostic Test: FDG-PET
- double negative group: patients with one type of PSMA-/FDG- homogeneous segment
  Interventions: Diagnostic Test: PSMA PET/CT scan; Diagnostic Test: FDG-PET
- PSMA predominant group: patients with one type of PSMA+/FDG- heterogeneous segment
  Interventions: Diagnostic Test: PSMA PET/CT scan; Diagnostic Test: FDG-PET
- FDG predominant group: patients with one type of PSMA-/FDG+ heterogeneous segment
  Interventions: Diagnostic Test: PSMA PET/CT scan; Diagnostic Test: FDG-PET

INTERVENTIONS:
Diagnostic Test: PSMA PET/CT scan — Different developing agents
Diagnostic Test: FDG-PET — Different developing agents

SUMMARY:
The purpose of this study is to analyze heterogeneity of prostate cancer（PCa）based on the head-to-head imaging of prostate-specific membrane antigen (PSMA) and fluorodeoxyglucose (FDG) positron emission tomography computed tomography (PET/CT)

DETAILED DESCRIPTION:
PET/CT examinations were performed on different days using Siemens Biograph MCT PET/CT equipment. All patients were examined on the same scanner. Patients were fasted for more than 6 h before [18F]FDG PET/CT examination, blood glucose was controlled below 11.1 mmol/L, [18F]FDG injection dose was 3.7 MBq/kg, and [18F]FDG PET/CT examination was performed after 60 min rest. [18F]PSMA-1007 injection dose was 3.7 MBq/kg, and PET/CT scan was performed 60 min after injection. To avoid interference of prostate lesion detection by active urine in the bladder, patients were asked to urinate or undergo forced diuresis before the start of the examination. The scan was performed from the top of the head to the base of the thighs. Low-dose CT was taken with automatic milliampere-second 120 kV voltage scans with a matrix of 512 × 512 and a thickness of 5 mm, and PET/CT image acquisition was taken from 5-6 beds for 2-3 min each. CT data was used for attenuation correction at the end of the acquisition, reconstructed by the two-iteration method (21 subsets in total), and the True X +TOF algorithm was applied to reconstruct the images. Two nuclear medicine physicians with extensive experience in PET/CT interpretation evaluated the images using the LIFEx software v 7.1.0. Both readers were blinded to both clinical and pathological data

ELIGIBILITY:
Inclusion Criteria:

* Untreated patients with PCa confirmed by prostate systemic pathological biopsy
* Patients underwent [18F]PSMA-1007 and [18F]FDG PET/CT and the imaging interval was less than one month.

Exclusion Criteria:

* Patients received treatment at intervals of two imaging
* Imaging was less than 1 week after pathology biopsy

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Subjects treated at the First Affiliated Hospital of China Medical University
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The relationship between imaging phenotypes and gleason score (GS) | From enrollment to the end of 1 month inspection

CONTACTS AND LOCATIONS:
Overall Officials: Xuena Li, PhD, Study Director — First Hospital of China Medical University
Locations (1):
- Department of Nuclear Medicine, The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided